CLINICAL TRIAL: NCT03403075
Title: Physical Therapy as "Drug, Non-drug"
Brief Title: Therapeutic Education in Physical Activity (ETAF)
Acronym: ETAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: GRADE Onlus (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAF2017
Record Dates: First submitted 2017-11-08; First posted 2018-01-18 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2020-01

CONDITIONS: Hematologic Neoplasms
Keywords: blood cancer; exercise; therapeutic education; fatigue; feasibility
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Control Group will be offered usual care (UC), plus two sessions of therapeutic education delivered in small groups. In these educational sessions, patients are provided with useful information on communication strategies, problem solving strategies, recognition and management of symptoms and the management of any aids/orthoses provided in everyday life, etc. In the meetings, it will be emphasized the importance of maintaining an active lifestyle as much as possible by encouraging involvement in physical activity even during the cancer treatment period.
  Written information material that summarizes the concepts addressed during group meetings will be provided.
  Interventions: Behavioral: Usual care
- ETAF: Therapeutic Education Physical Activity (Experimental): Intervention group will perform UC, and the two sessions of therapeutic education delivered in small group, as for the Control Group. The Intervention group will also provided for 6 individual sessions of therapeutic education and physical activity held by physiotherapists dedicated to the study, according to the patients' needs and objectives.
  In these sessions, the topics discussed in group will be deepened, personalizing them according to the patient's characteristics. Furthermore, personalized physical activity is planned, taking into account the context of execution, the clinical condition and the patient's preferences. The patient will be trained to build an action plan aimed at self-plan physical activities and a diary will be provided to monitor the physical activity carried out autonomously.
  Written information material that summarizes the concepts addressed during group and individual sessions will be provided.
  Interventions: Behavioral: ETAF

INTERVENTIONS:
Behavioral: ETAF — Therapeutic education and Physical activity
  Arms: ETAF: Therapeutic Education Physical Activity
Behavioral: Usual care — Usual care
  Arms: Usual Care

SUMMARY:
To date, studies published on multidimensional rehabilitation programs are addressed to patients with different types of cancer and, frequently, these studies only include a limited number of patients with blood neoplasms. So, there is no evidence of the effectiveness of multidimensional rehabilitation programs in this particular category of patients. A systematic review of the effectiveness of aerobic exercise alone, not associated with therapeutic education, has recently been conducted in adult individuals with hematological malignancies (reference 25386666). The review highlighted the effectiveness of physical activity on the quality of life of the target population. However, the medium and long term effects that physical exercise have on other clinically relevant endpoints, such as fatigue, psychological distress, and physical performance level, remain to be clarified. Thus, it is important to investigate the effectiveness of multidimensional interventions that integrate physical activity to therapeutic education targeted at the specific needs of individuals with blood neoplasm.

The aim of this study is to evaluate, in blood cancer patients, the feasibility of a therapeutic education program associated with physical activity, and to verify its effect by a long-term follow-up.

DETAILED DESCRIPTION:
This is a randomized controlled pilot study • Control Group will be offered usual care (UC), which includes two sessions of therapeutic education delivered in small groups. In these educational sessions, patients are provided with useful information on communication strategies, problem solving strategies, recognition and management of symptoms and the management of any aids/orthoses provided in everyday life, etc. In the meetings, it will be emphasized the importance of maintaining an active lifestyle as much as possible by encouraging involvement in physical activity even during the cancer treatment period.

Written information material that summarizes the concepts addressed during group meetings will be provided.

• Intervention group will be offered therapeutic education as described for the control group, plus 6 individual sessions of therapeutic education and physical activity (ETAF). The 6 individual session will be held by a physiotherapist dedicated to the study, on a weekly / bi-weekly basis, according to the objectives set and the needs of the patient.

In these sessions, the topics already discussed in group will be deepened, personalizing them according to the patient's characteristics. Furthermore, personalized physical activity is planned, taking into account the context of execution, the clinical condition and the patient's preferences. Patients will be trained to build an action plan aimed at self-plan physical activities and a diary will be provided to monitor the physical activity carried out autonomously.

Written information material that summarizes the concepts addressed during group and individual sessions will be provided.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of blood cancer or early relapse of blood cancer

Exclusion Criteria:

* Expected prognosis <12 months
* Clinical or anamnestic conditions preventing participation in the rehabilitation program (dementia, non-collaboration for major psychiatric disorders, blindness, deafness, any language barriers or communication deficits that prevent participation in the program, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to ETAF | 18 months (on average) - through study completion
  rate of adherence to experimental intervention: ratio between planned intervention and actual intervention (process indicator).

SECONDARY OUTCOMES:
Effect size on Fatigue | 6 months
  The size of the effect of ETAF, compared to the usual care, will be estimated on cancer-related fatigue (FACIT Fatigue Scale);
Effect size on QoL | 6 months
  The size of the effect of ETAF, compared to the usual care, will also be estimated on quality of life (EORTC Quality of life Questionnaire-C30);
Effect size Psychological distress | 6 months
  The size of the effect of ETAF, compared to the usual care, will also be estimated on psychological distress (NCCN Distress Thermometer and Problem list for patients);
Effect size on Physical function | 6 months
  The size of the effect of ETAF, compared to the usual care, will also be estimated on Physical function (Time up and go and 6MWT)

OTHER OUTCOMES:
Effect of patient education - adherence | 6 months
  The effect of the educational intervention will be assessed through:
  - degree of patient's adherence to an active lifestyle (Kirkpatrick's taxonomy level 4) (Kirkpatrick, 1996).
Effect of patient education - satisfaction | 6 months
  The effect of the educational intervention will be assessed through:
  - degree of satisfaction of the patient involved in the study and perception of the utility of the treatment provided (Kirkpatrick's taxonomy level 1) (Kirkpatrick, 1996).

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, MD, Principal Investigator — AUSL - IRCCS of Reggio Emilia; Stefania Costi, PT, Study Chair — AUSL - IRCCS of Reggio Emilia and University of Modena and Reggio Emilia
Locations (1):
- Local Health Authority - IRCCS of Reggio Emilia, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergenthal N, Will A, Streckmann F, Wolkewitz KD, Monsef I, Engert A, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2014 Nov 11;(11):CD009075. doi: 10.1002/14651858.CD009075.pub2. PMID 25386666
- [Background] Kirkpatrick, DL. Great ideas revisited: revisiting Kirkpatrick's four-level model. Training and Development. 1996; 50:54-58.
- [Derived] Accogli MA, Denti M, Costi S, Fugazzaro S. Therapeutic education and physical activity are feasible and safe in hematologic cancer patients referred to chemotherapy: results of a randomized controlled trial. Support Care Cancer. 2022 Dec 19;31(1):61. doi: 10.1007/s00520-022-07530-4. PMID 36534365
- [Derived] Denti M, Accogli MA, Costi S, Fugazzaro S. Therapeutic Education and Physical Activity to Support Self-management of Cancer-related Fatigue in Hematologic Cancer Patients: Protocol of a Feasibility Randomized Controlled Trial. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420969830. doi: 10.1177/1534735420969830. PMID 33243016